CLINICAL TRIAL: NCT03625388
Title: Randomized, Open-Label, Phase II, Multicenter, Multi-Country Study to Evaluate Safety and Efficacy of Dasatinib 50 mg in First-Line Treatment of Early Chronic Phase Chronic Myeloid Leukemia
Brief Title: Low Dose Dasatinib (50 mg Daily) as First-line Treatment for Newly Diagnosed Chronic-Phase Chronic Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hikma Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPI-JOR-LEB-KSA-TUN-2017-01
Record Dates: First submitted 2018-08-02; First posted 2018-08-10 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: Leukemia, Myeloid, Philadelphia Positive; Dasatinib; Generic Dasatinib; Dasatinib 50 mg once daily; Early chronic phase chronic myeloid leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — Dasatinib; elsulfavirine

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized to receive either dasatinib 50 mg or dasatinib 100 mg orally once daily for the duration of the study which is 18 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dasatinib 50 mg (Other): Dasatinib 50 mg orally once daily
  Interventions: Drug: Dasatinib
- Dasatinib 100 mg (Other): Dasatinib 100 mg orally once daily
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Film coated tablet contains dasatinib monohydrate
  Other Names: Elpida®

SUMMARY:
The purpose of this multicenter randomized study is to compare efficacy and safety of dasatinib 50 mg once daily and dasatinib 100 mg once daily in patients with early chronic phase (CP) chronic myeloid leukemia (CML)

DETAILED DESCRIPTION:
A multicenter, prospective, open-label, randomized Phase II study to compare efficacy by measuring rates of major molecular response (MMR) at 12 months in patients with Ph+ chronic phase (CP) chronic myeloid leukemia (CML) randomized to receive either dasatinib 50 mg QD or dasatinib 100 mg QD. Approximately 100 patients are expected to be randomized. The duration of patient participation will be 18 months

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Diagnosis of Ph+ or BCR-ABL positive CML in early CP (i.e. time from diagnosis <12 months). Except for hydroxyurea and/or 1-2 doses of cytarabine (up to 6g/m2 total), patients must have received no or minimal prior therapy, defined as 30 days of prior approved tyrosine kinase inhibitor (TKI).
3. Clonal evolution defined as the presence of additional chromosomal abnormalities other than the Ph-chromosome has been historically included as a criterion of accelerated phase (AP). However, patients with clonal evolution as the only criterion of AP have a significantly better prognosis, and when present at diagnosis may not impact the prognosis at all. Thus, patients with clonal evolution and no other criteria for AP will be eligible for this study.
4. ECOG performance of 0-2.
5. Adequate end organ function defined as the following: total bilirubin <1.5x ULN (unless secondary to Gilbert's disease, in which case it should be <2.5x ULN), SGPT <2.5x ULN, creatinine <1.5x ULN.
6. Patients must sign an informed consent form (ICF) indicating they are aware of the investigational nature of this study, in keeping with the policies of the hospital

Exclusion Criteria:

1. NYHA cardiac class 3-4 heart disease
2. Cardiac symptoms - Patients meeting the following criteria are not eligible unless cleared by a cardiologist:

   1. Uncontrolled angina within 3 months
   2. Diagnosed or suspected congenital long QT syndrome
   3. Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
   4. Prolonged QTc interval on pre-entry electrocardiogram (>460 msec)
3. History of significant bleeding disorder unrelated to cancer including:

   1. Diagnosed congenital bleeding disorders (e.g. Von Willebrand's disease)
   2. Diagnosed acquired bleeding disorder within one year (e.g. acquired anti-factor VIII antibodies)
   3. Isolated thrombocytopenia without recurrent bleeding episodes shall be considered eligible for study entry
4. Patients with active uncontrolled psychiatric disorders including: psychosis, major depression, and bipolar disorders
5. Women of pregnancy potential must practice an effective method of birth control, unless otherwise instructed, during the course of the study in a manner such that risk of failure is minimized

   1. Prior to study enrollment, women of childbearing potential (WOCBP) must be advised of the importance of avoiding pregnancy during study participation and the potential risk factors for an unintentional pregnancy
   2. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential
   3. Women must continue birth control for the duration of the study and at least 3 months after the last dose of study drug
6. Pregnant or breast-feeding women are excluded

   a. All WOCBP must have a negative pregnancy test prior to first receiving the study drug. If the pregnancy test is positive, the patient must not receive the study drug and must not be enrolled in the study.
7. Patients in late chronic phase (i.e. time from diagnosis to treatment >12 months), accelerated phase (except as noted in inclusion criteria 2) or blast phase are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2023-07-22 (Actual); Study Completion 2023-07-22 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who achieve and maintain MMR at 12 months using RQ-PCR test | 12 months
  Major molecular response (MMR) is defined as BCR-ABL1 ≤ 0.1%

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) to dasatinib | 18 months
  Evaluation of adverse events (AEs), serious AEs (SAEs), and clinically relevant changes in laboratory tests according to laboratory reference ranges
Transformation free survival (TFS) in eligible patients randomized to dasatinib 50 mg or dasatinib 100 mg treatment arms | 18 months
  Transformation free survival was measured from the start of therapy to the date of transformation to accelerated or blastic phases while on therapy or to the date of last follow-up.
Event free survival (EFS) | 18 months
  EFS is measured from the start of treatment to the date of any of the following events : loss of CHR, loss of CCyR or MCyR, dose escalation, discontinuation of therapy for toxicity or lack of efficacy, progression to AP or BP, or death from any cause at any time
Blastic phase (BP) transformation | 18 months
  BP is defined as the presence of 30% blasts or more in the peripheral blood or bone marrow
Overall survival | 18 months
  Overall survival time is defined as the time from date of randomization until the date of death from any cause at any time or date of last follow up
Proportion of patients with Complete cytogenetic response (CCyR) at 12 months | 12 months
  defined as 0% Ph+ metaphases, or FISH ≤2%, or BCR-ABL transcripts (IS) ≤1%
Proportion of patients with MR 4.5 at 18 months | 18 months
  (BCR-ABL transcripts ≤ 0.0032%)
Health-Related Quality of Life (HRQoL): EORTC QOLCML24 | 18 months
  Mean change in Health-Related Quality of Life (HRQoL) utilizing EORTC QOLCML24 questionnaire throughout treatment visits
Frequency of not taking the medications as prescribed | 18 months
  Evaluated by identifying the frequency of not taking the medications as prescribed and the reasons. The decision on non-compliance is based on the treating physician's judgment.

CONTACTS AND LOCATIONS:
Locations (5):
- Jordan (2):
  - King Hussein Cancer Center (KHCC), Amman
  - Jordan University Hospital (JUH), Amman
- American University of Beirut Medical Center (AUBMC), Beirut, Lebanon
- The King Faisal Specialist Hospital and Research Centre (KFSH&RC), Riyadh, Saudi Arabia
- Aziza Othmana Hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No